CLINICAL TRIAL: NCT00456482
Title: A Multicenter, Randomized, Double-Masked, Controlled Study to Evaluate the Safety and Efficacy of an Intravitreal Fluocinolone Acetonide Implant in Subjects With Non-Infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy of Fluocinolone Acetonide Intravitreal Implant
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: SARS epidemic in Asia and Canada
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 415-004
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Non-infectious Uveitis
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluocinolone Acetonide 0.59mg (Experimental): Fluocinolone acetonide intravitreal implant 0.59mg
  Interventions: Drug: Fluocinolone Acetonide 0.59mg
- Fluocinolone Acetonide 2.1mg (Experimental): Fluocinolone acetonide intravitreal implant 2.1mg
  Interventions: Drug: Fluocinolone Acetonide 2.1mg
- No Intervention (No Intervention): Fellow eye

INTERVENTIONS:
Drug: Fluocinolone Acetonide 0.59mg — Fluocinolone Acetonide Intravitreal Implant 0.59 mg
  Arms: Fluocinolone Acetonide 0.59mg
Drug: Fluocinolone Acetonide 2.1mg — Fluocinolone Acetonide Intravitreal Implant 2.1 mg
  Arms: Fluocinolone Acetonide 2.1mg

SUMMARY:
This is a multi-center, randomized, double-masked, controlled study to evaluate the safety and efficacy of fluocinolone acetonide intravitreal implants for the management of subjects with non-infectious uveitis affecting the posterior segment of the eye. An additional objective is to compare the safety and efficacy of two doses of fluocinolone acetonide.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females at least 6 years of age who had been diagnosed and treated for recurrent,
* Non-infectious uveitis affecting the posterior segment of one or both eyes for at least 1 year prior to the start of the study,
* Had clinically 'quiet' eyes at surgery.

Exclusion Criteria:

* Coexistent medical or ocular conditions that would interfere with obtaining or interpreting data for this study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2002-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of uveitis before and after implantation. Postimplantation recurrences were evaluated using protocol-defined criteria based upon changes in VA, vitreous haze, and the presence of cells in the anterior chamber of the eye. | 1 year pre-implantation; 3 years post-implantation

SECONDARY OUTCOMES:
Between-dose group and within-subject comparisons (Study to Fellow eye) for uveitis recurrence; time to first recurrence; need for adjunctive uveitis treatment; reduction in the area of cystoid macular edema; results of quality of life surveys. | 1 year pre-implantation; 3 years post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Comstock, OD, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Background] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128